CLINICAL TRIAL: NCT01443000
Title: Survey of Patients With Idiopathic Orbital Inflammation Syndrome (IOIS): Clinical, Morphological and Pathological Features and Treatment Outcomes
Brief Title: Survey of Patients With Idiopathic Orbital Inflammation Syndrome
Acronym: SIOI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI08014; 2010-A00512-37 (Other: IDRCB)
Record Dates: First submitted 2011-06-15; First posted 2011-09-29 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Orbital Ischemic Syndrome; Orbital Pseudotumor
Keywords: Observational study; IOIS; Orbital Pseudotumor; Outcome; Treatment
MeSH Terms: conditions — Orbital Pseudotumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be frozen to form a serum storage and a DNAthèque. These samples will achieve further analysis based on the evolution of knowledge on mechanisms contributing to the orbital inflammation.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterise the clinical features, histopathology and the treatment outcomes of patients with idiopathic orbital inflammation syndrome.

DETAILED DESCRIPTION:
Idiopathic orbital inflammatory syndrome (IOIS) is a heterogeneous group of disorders characterised by orbital inflammation without any identifiable local or systemic causes. It is a rare clinical entity and a diagnosis of exclusion. Lymphomas, thyroid eye diseases or systemic diseases can have similar presentation and so, a histopathological diagnosis is considered important. IOIS is a difficult condition to treat. Compilation of reported small series of patients with IOIS suggested that they require multiple systemic immunosuppressant drugs and radiotherapy. Recently, a large monocentric study including patients with biopsy proven IOIS showed that up to 40% of them can relapse. Their clinical and pathological features did not correlate with treatments outcomes. The investigators decide therefore to conduct a multicentric retro/ prospective study to determine clinical features, histopathology and treatment outcomes of French patients with IOIS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven IOIS or presumed IOIS
* Patients with chronic IOS
* Patient with inaugural IOIS or being treated for IOIS

Exclusion Criteria:

* Patients who do not fulfill the inclusion criteria
* Patients with systemic disease-associated IOIS
* Incomplete follow-up of patients treated for IOIS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for IOIS
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2012-03-03 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of remission, relapse or resistance among patients with IOIS during the 24 month follow-up | The remission, relapse, or the resistance at inclusion (for those previously diagnosed as IOIS), and at 6, 12, 18 and 24 months
  Remission: absence of steroids, their withdrawal or their pursuit at a dose ≤ 10 mg/d in the absence of immunosuppressor treatment.
  Relapse: re initiation of steroids, or their ascension in patients for whom they have been reduced to less than 20 mg/d.
  Resistance: inability to reduce steroids at an effective dose ≤ 20 mg/d.

SECONDARY OUTCOMES:
Histopathological classification of IOIS patients | at diagnostic
  -Histopathological forms of the IOIS patients at diagnosis, according to the classification described by Mombaerts, namely: classical orbital pseudotumor, sclerosing orbital pseudotumor, granulomatous orbital pseudotumor and vasculitic pseudotumor.
Ophthalmologic features (laterality, pain, visual acuity, eye movement and eyelid) | at diagnosis and in case of remission, or relapse, or resistance
  The clinical manifestations of systemic diseases mentioned below, will be evaluated in case of relapse or resistance: Grave's disease or auto immune thyroiditis, sarcoidosis, Wegener's granulomatosis, polyarteritis nodosa, Churg- Strauss syndrome, systemic lupus erythematosus and Gougerot-Sjögren syndrome.
MRI features (muscle enlargement, irregular borders, extension to the orbital fat, enhancement around globe) of patients with IOIS | at diagnosis and in case of remission, or relapse, or resistance.
  the lesional topography and the T1/T2 weighted sequences will be studied
Immunologic features of IOIS patients | at inclusion
  the IgG4 level and ANA in sera will be assessed
Cumulated dose of prednisone | at remission, or relapse, or resistance
Incidence of orbital lymphomas | at 6, 12, 18, 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien ABAD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine interne - Hôpital Avicenne, Bobigny, France